CLINICAL TRIAL: NCT07201779
Title: Reducing Emotional Distress for Childhood Hypoglycemia in Parents (REDCHiP) -A Feasibility Randomized Controlled Trial in the Portuguese Context
Brief Title: Adaptation of REDCHIP Intervention for the Portuguese Context
Acronym: REDCHIP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ISPA - Instituto Universitario de Ciencias Psicologicas, Sociais e da Vida (Other)
Collaborators: Hospital de Santa Maria, Portugal (Other); Hospital Dona Estefânia, Centro Hospitalar de Lisboa Central, Lisboa (Unknown); Fundação para a Ciência e a Tecnologia (Other); Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Vasco Vicente Costa, Principal Investigator, ISPA - Instituto Universitario de Ciencias Psicologicas, Sociais e da Vida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 114/24 and Inv 631
Record Dates: First submitted 2025-09-22; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes
Keywords: REDCHiP; Portuguese Context; Protocol; Psychological Interventions; Parents; Young Children; Type 1 Diabetes; Telehealth
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REDCHIP Intervention Group (Experimental): REDCHIP intervention group will receive 10 telehealth group sessions. CBT strategies are utilized to increase parents' awareness of any maladaptive thoughts and behaviors they may have related to FH (e.g., fear associated with in target glucose levels, reducing insulin to maintain higher glucose levels) and help them to adopt more adaptive coping skills. REDCHiP also includes content to improve participant's parenting skills and some T1D education to promote parents' knowledge and skills related to managing their young child's T1D
  Interventions: Behavioral: REDCHiP
- Treatment As Usual Control Group (Active Comparator): These participants will receive the usual treatment provided during their medical appointments
  Interventions: Other: Treatment As Usual Control Group

INTERVENTIONS:
Behavioral: REDCHiP — REDCHIP comprises 10 telehealth group sessions for parents of young children with T1D, is grounded in Cognitive Behavioral Therapy (CBT) principles, and is designed to address parents FH, and their avoidant coping behaviors related to FH. Sessions also focus on strengthening parents' coping strategies associated with T1D management and helping them to reduce feelings of diabetes distress.
  Arms: REDCHIP Intervention Group
Other: Treatment As Usual Control Group — Participants will receive their treatment as usual in medical appointments
  Arms: Treatment As Usual Control Group

SUMMARY:
The present Feasibility Randomized Controlled Trial (FRCT) aims to assess the acceptability and effectiveness of REDCHiP intervention, targeting parents of young children with T1D, followed in two major Portuguese hospitals. The objective of this trial is to evaluate (1) acceptability and feasibility by evaluating recruitment and retention rates, attendance throughout the sessions, and responses to parent satisfaction; (2) effectiveness by analyzing changes in parents' FH, diabetes distress (DD), emotional regulation (ER), resilient coping skills (RC), and anxiety and depression as well as changes in child glycemic outcomes (HbA1c, GMI, TBR, TIR, TAR) at three time points among participants allocated on intervention versus Treatment As Usual (TAU) group. Finally, (3) the investigators aim to qualitatively evaluate participant´s experiences and feedback regarding the REDHIP intervention through interviews.

DETAILED DESCRIPTION:
One of the principal fears experienced by parents of young children with T1D is related to the occurrence of hypoglycemia episodes. These events can occur on a daily basis (i.e., often triggered by excessive exercise and/or prolonged periods without food intake) and can lead to severe acute consequences (i.e., seizures and coma) as well as long-term complications (i.e., cognitive decline). Moreover, young children often demonstrate reduced awareness for hypoglycemia and a limited ability to report its symptoms (i.e., sweating, shaking and dizziness) making it challenging for parents and other adult caregivers to detect and treat a hypoglycemic event. Combined these circumstances significantly contribute to heightened parental FH, which in some cases escalate into clinical phobia. In line with the theoretical model of caregiver fear of hypoglycemia, higher parental FH is frequently associated with avoidant behaviors and maladaptive coping strategies related to hypoglycemia. These patterns may contribute to persistently higher glycemic levels and increased variability, which, in turn, can serve as a catalyst for the development of T1D complications in their child. The literature has highlighted the potential impact of parental FH on children's glycemic outcomes and T1D management. It is also unclear whether routine use of an insulin pump or continuous glucose monitor can help to reduce FH in parents of very young children with T1D without the addition of psychological support, suggesting it is a high priority to design and test interventions to effectively treat parental FH, enhance parental well-being, and promote their T1D treatment engagement.

Thus, the original structure of the manualized REDCHiP intervention, is 10 video-based telehealth sessions (i.e.,7 group and 3 individual sessions with duration of 30 to 60 minutes). The present format of the Portuguese REDCHiP will have a 10 video-based telehealth sessions, all in group format, targeting parents of young children (≤ 8 years old) with T1D followed on two major hospitals in Lisbon, Portugal (i.e., Santa Maria Hospital and Dona Estefânia Hospital). This intervention is grounded in Cognitive Behavioral Therapy (CBT) principles, and is designed to address parents FH, and their avoidant coping behaviors related to FH. In addition, the sessions also focus on strengthening parents' coping strategies associated with T1D management and helping them to reduce feelings of diabetes distress Based on previous REDCHiP findings, and with the reported acceptability and feasibility of the intervention study, the investigators hypothesize that participants of intervention group will report lower levels of FH and better glycemic outcomes at immediate post-intervention compared to TAU group. The investigators anticipate group differences in these outcomes at three-month follow up. Furthermore, the investigators expect that REDCHiP will lead to improvements in all psychosocial adjustment factors (i.e., FH, DD, ER, RC, anxiety and depression) among all parents after receiving the REDCHiP intervention.

Accordingly, this protocol outlines the first attempt to culturally adapt and implement the telehealth REDCHiP intervention beyond the United States context.

ELIGIBILITY:
Inclusion Criteria:

1. Primary caregivers must have a young child aged ≤ 8 years with a confirmed diagnosis of T1D for at least three months;
2. Young children must be using either an continuous subcutaneous insulin infusion (CSII) or multiple daily insulin injections (MDI) and continuous glucose monitoring (CGM) for daily T1D treatment;
3. Parents must have internet access and a computer, tablet or smartphone that connects to the internet.

Exclusion Criteria:

1. Parents with severe psychiatric diagnosis;
2. Families of children with another severe chronic condition (e.g., chronic kidney disease and Crohn's disease);
3. Parents who are not fluent in Portuguese.

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Parents Fear of Hypoglycemia | From baseline to post-intervention (14-15 week)
  Parents Fear of Hypoglycemia will be collected trough: The Hypoglycemia Fear Survey - Parents (HFS-P), 18-item self-report measure and comprises a total score and two subscales: Behavior and Worry.
Parents Diabetes Distress | From baseline to post-intervention (14-15 week)
  Parents Diabetes Distress will be evaluated by, Parents The Problem Areas in Diabetes - Parent Revised (PAID-PR), 18-item self-report measure. It comprises two subscales: Immediate Burden and Theoretical Burden.
Children Glycemic Outcomes | From baseline to post-intervention (14-15 week)
  Children´s Glycated Hemoglobin (HbA1c)
Children Glycemic Outcomes | From baseline to post-intervention (14-15 week)
  Time in Range (TIR)
Children Glycemic Outcomes | From baseline to post-intervention (14-15 week)
  Glucose Management Indicator (GMI)
Children Glycemic Outcomes | From baseline to post-intervention (14-15 week)
  Time Bellow Range (TBR)
Children Glycemic Outcomes | From baseline to post-intervention (14-15 week)
  Time Above Range (TAR)

CONTACTS AND LOCATIONS:
Overall Officials: Vasco V Costa, MD, Principal Investigator — William James Center for Research (ISPA)

IPD SHARING:
Plan to Share IPD: No